CLINICAL TRIAL: NCT05495334
Title: Innovations in Genicular Outcomes Registry
Acronym: iGOR
Status: Recruiting | Type: Observational
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IOV-REG-001
Record Dates: First submitted 2022-07-14; First posted 2022-08-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All participants: Eligible and enrolled subjects with knee OA pain who require treatment on the target knee as a part of pain management.
  Interventions: Procedure: Treatment for Knee OA

INTERVENTIONS:
Procedure: Treatment for Knee OA — Pain management treatment for knee OA.

SUMMARY:
The registry will capture prospective data on patients receiving pain management for chronic pain due to knee osteoarthritis (OA) or pain optimization for knee arthroplasty due to knee OA. The OA pain therapies may include cryo nerve block, radiofrequency ablation (RFA), intra-articular (IA) corticosteroids, viscosupplementation, opioids, and others (e.g., non-steroidal anti-inflammatory drugs [NSAIDs]).

ELIGIBILITY:
Inclusion Criteria:

1. Planned to receive treatment for knee OA pain including, but not limited to, knee injections, nerve blocking procedures, or knee arthroplasty within 60 days of screening
2. Able to understand the informed consent and assessment questionnaires and have the ability to complete them in the opinion of the investigator
3. Have access to a smartphone or internet access with a computer/tablet to complete the questionnaires using the registry application

Exclusion Criteria:

1. Actively enrolled in an investigational trial that would preclude patients from receiving the site's standard of care for knee OA pain or knee arthroplasty recovery protocol
2. Planning to have a surgery other than on the target knee

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are planned to receive treatment within 60 days of screening for knee OA pain will be screened, and if eligible, will be approached for participation in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and interference scores via NRS (Numeric Rating Scale) | 18 months
  NRS score from 0(being none)-10(being the worst)
Pain intensity and interference scores via BPI-sf (Brief Pain Inventory-short form) | 18 months
  Pain intensity and interference scores via BPI-sf 0 to 10, where: 0 = no pain and 10 = pain as bad as you can imagine
Opioid use via pre-and post-treatment analgesic medication use log | 18 months
  Opioid use via pre-and post-treatment analgesic medication use log
Functional status via KOOS-JR (Knee injury and Osteoarthritis Outcome Score for Joint Replacement) | 18 months
  Functional status via KOOS-JR. 0(none)-4(extreme)
Functional status via SANE (Single Assessment Numeric Evaluation) | 18 months
  Functional status via SANE. Percentage of normal (0% to 100% scale with 100% being normal)
Quality of Sleep via PROMIS-SD (PROMIS - Sleep Disturbance - Short Form 8b) | 18 months
  Quality of Sleep via PROMIS-SD. 1(Best)-5(Worst)
Adverse events related to pain therapies | 18 months
  Adverse events related to pain therapies
General HRQOL via PROMIS-10 (PROMIS GLOBAL-10) | 18 months
  General HRQOL via PROMIS-10. 1(Best)-5(Worst)
Patient Satisfaction | 18 months
  Patient satisfaction with pain management questionnaire (Patient Satisfaction Questionnaire). Two questions assessing satisfaction and benefit.
Physical therapy utilization and work productivity via PT/Work Productivity | 18 months
  Physical therapy (PT) utilization and work productivity via PT/Work Productivity (WP) questionnaire.
Emergency Department (ED) visits | 18 months
  Emergency Department (ED) visits
Reimbursement status | 18 months
  Reimbursement status
Post-operative pain scores NRS (Numeric Rating Scale) | 18 months
  Post-operative pain scores (NRS) 0(being none)-10(being the worst)
Post-operative opioid consumption (analgesic medication use log) | 18 months
  Post-operative opioid consumption (analgesic medication use log)
Length of facility stay | 18 months
  Length of facility stay

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - The MORE Foundation, Phoenix, Arizona
  - Orthopedic Education and Research Institute of So Ca (Hoag), Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - MidState Orthopedics and Sports Medicine, Alexandria, Louisiana
  - Louisiana State University /Ochsner, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Henry M Jackson Foundation for the Advancement of Military Medicine/Walter Reed National Military Medical Center, Bethesda, Maryland
  - OrthoNebraska Clinics, Omaha, Nebraska
  - Jersey City Medical Center, Jersey City, New Jersey
  - Northwell Health, Garden City, New York
  - Genesee Orthopedics and Plastic Surgery (St. Elizabeth Med Center/ Apex Surgical Center), New Hartford, New York
  - Blue Nine Systems, Asheville, North Carolina
  - Oklahoma Surgical Hospital, Tulsa, Oklahoma
  - Penn Highlands DuBois, DuBois, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasa V, Mihalko W, Rivadeneyra A, Urban J, Wickline A, Rogenmoser D, Concoff A, Spitzer A, Mont MA. Innovations in Genicular Outcomes Registry (IGOR): protocol for a real-world registry study of treatments for knee osteoarthritis. Ther Adv Musculoskelet Dis. 2024 Dec 16;16:1759720X241304193. doi: 10.1177/1759720X241304193. eCollection 2024. PMID 39691173